CLINICAL TRIAL: NCT03159819
Title: Clinical Study of Redirected Autologous T Cells With a Claudin18.2-targeted Chimeric Antigen Receptor in Patients With Advanced Gastric Adenocarcinoma and Pancreatic Adenocarcinoma
Brief Title: Clinical Study of CAR-CLD18 T Cells in Patients With Advanced Gastric Adenocarcinoma and Pancreatic Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Bin Wang, Attending physician, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG4003
Record Dates: First submitted 2017-05-11; First posted 2017-05-19 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Advanced Gastric Adenocarcinoma; Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-CLD18 T cells (Experimental): Autologous T Cells with a Claudin18.2-redirected Chimeric Antigen Receptor. Route of administration: Intravenous injection.
  Lymphodepletion conditioning regimen will be applied prior to CAR-CLD18 T cell infusion.
  Interventions: Genetic: CAR-CLD18 T Cells

INTERVENTIONS:
Genetic: CAR-CLD18 T Cells — Dose escalation will be applied in this study.
  Other Names: Claudin18.2-redirected Autologous Cells

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety, tolerability and engraftment of CAR-CLD18 T cells in patients with advanced gastric adenocarcinoma and pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
For patients with gastric adenocarcinoma who have not been cured with first line chemotherapy, and who are not willing to undergo second line chemotherapy after the failure of first line chemotherapy while there are no effective therapies for their unmet medical needs known at this time, and for patients with advanced/metastatic pancreatic adenocarcinoma which has relapsed after surgery or for which there is no surgical indication, who have not been cured with or refused to receive other standard regimens, single or multiple doses of CAR-CLD18 T cells will be given to observe safety and efficacy of CAR-CLD18 T cells.

Primary objectives:

Determine the safety, tolerability and cytokinetics of the autologous T cells transduced with anti-Claudin18.2 lentiviral vector in patients with gastric adenocarcinoma and pancreatic adenocarcinoma.

Secondary objectives:

Make a preliminary evaluation on the efficacy of CAR-CLD18 T cells in patients with gastric adenocarcinoma and pancreatic adenocarcinoma with the following parameters:

Time of tumor progression (TTP);

Disease Control Rate (DCR);

Objective Remission Rate (ORR);

Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 - 70 with pathologically confirmed advanced gastric adenocarcinoma and pancreatic adenocarcinoma.
2. Biopsy confirmation of Claudin18.2 positive.
3. Patients with advanced gastric adenocarcinoma who have not been cured with second line chemotherapy, and who are not willing to undergo second line chemotherapy after the failure of first line chemotherapy. (1) Failure of treatment is defined as disease progression, recurrence or metastatic disease, or intolerable toxicities occurred after treatment. (2) Each line of treatment during the period of disease progression includes one or more chemotherapy drugs which are administered for not less than one cycle or even longer. Neoadjuvant/adjuvant therapy can be applied at an earlier stage of treatment. If patient has developed recurrence or metastatic disease within 24 weeks of neoadjuvant/adjuvant therapy, it is considered as one line of systemic chemotherapy. (3) Therapies that can be performed at an earlier stage are chemotherapy in conjunction with molecular targeted drugs.
4. Patients with advanced/metastatic pancreatic adenocarcinoma which has relapsed after surgery or for which there is no surgical indication, who have not been cured with or refused to receive other standard regimens.
5. Expected survival after first dose of study drug > 12 weeks.
6. At least one measurable lesion (≥ 10 mm) for imaging assessment.
7. ECOG scores 0 - 1.
8. Adequate venous access for apheresis and venous blood sampling, and no other contraindications for leukapheresis.
9. White blood cells (WBCs) ≥ 2.5×10^9/L Platelets (PLT) ≥ 100×10^9/L Hemoglobin, Blood (Hb) ≥ 9.0 g/dL MID ≥ 1.5×10^9/L Lymphocyte (LY) ≥ 0.47×10^9/L LY% ≥ 15%
10. Serum albumin (Alb) ≥ 30 g/L
11. Serum lipase (LPS) and serum amylase < 1.5 ULN
12. Serum creatinine ≤ 1.5 ULN
13. Alanine aminotransferase (ALT) ≤ 2.5 ULN Aspartate aminotransferase (AST) ≤ 2.5 ULN If osseous metastasis or liver metastasis is developed and alkaline phosphatase (ALP) > 2.5 ULN, ALT and AST < 1.5 ULN.
14. Serum total bilirubin (TBIL) ≤ 1.5 ULN
15. Prothrombin Time (PT): International Normalized Ratio (INR) < 1.7. PT < (ULN + 4) s

All test results should be within their normal ranges, and the patient is not receiving continuous supportive care.

Exclusion Criteria:

* Patients with any of the following conditions are not eligible for the study.

  1. Pregnant or lactating women.
  2. HIV positive, HCV positive, HBV DNA copies ≥ 10^3.
  3. Uncontrolled active infection.
  4. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
  5. Allergic to immunotherapies and related drugs.
  6. Untreated brain metastases or having symptoms of brain metastases.
  7. Metastases to the lung: central tumor or multiple metastases.
  8. Patients with heart disease for which treatment is needed or with poorly controlled hypertension.
  9. Patients with unstable or active peptic ulcer or with alimentary tract hemorrhage.
  10. Patients with previous organ transplantation or in preparation for organ transplantation.
  11. Patients in need of anticoagulant treatment (e.g. warfarin or heparin).
  12. Patients in need of long-term antiplatelet treatment (aspirin, dosage > 300 mg/d; clopidogrel, dosage > 75 mg/d).
  13. Previous treatment with chemoradiotherapy and tumor-targeting drug which were conducted 4 weeks prior to the study (blood collection).
  14. Patients have undertaken major surgeries or have been badly injured 4 weeks before the study (blood collection), or will undertake major surgeries during the study.
  15. The judgment of investigators that the patient is not able to or not willing to follow the instructions of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance | 24 weeks
  During the trial conduction, especially within the 24 weeks of treatment phase when CAR-CLD18 T cell administered, all adverse events (including laboratory abnormality and clinical events) will be closely monitored, and all ≥ grade 3 adverse events per CTCAE (v 3.0) will be recorded, including but not limited to the toxicities potentially suspected to relate to infusion procedures and/or CAR-CLD18 T cell therapy as listed below:
  * Fever
  * Chills
  * Nausea, vomiting and other gastrointestinal symptoms
  * Fatigue
  * Hypotension
  * Respiratory distress
  * Tumor lysis syndrome
  * Cytokine release syndrome
  * Neutropenia, thrombocytopenia
  * Liver and kidney dysfunction

SECONDARY OUTCOMES:
Engraftment | 2 years
  Duration of in vivo survival of CAR-CLD18 T cells is defined as "engraftment". The primary engraftment endpoint is the number of DNA vector copies per mL blood of CAR-CLD18 T cells at regular intervals through week 4 following the initial infusion. Q-PCR for CAR-CLD18 T vector sequences will be performed until any 2 sequential tests are negative, documented as engraftment and persistence of CAR-CLD18 T cells.

OTHER OUTCOMES:
Anti-tumor responses to CAR-CLD18 T cell infusions | 2 years
  Disease Control Rate (DCR)
Anti-tumor responses to CAR-CLD18 T cell infusions | 2 years
  Progression-free Survival (PFS)
Anti-tumor responses to CAR-CLD18 T cell infusions | 2 years
  Time of Tumor Progression (TTP)
Anti-tumor responses to CAR-CLD18 T cell infusions | 2 years
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Xianbao Zhan, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided